CLINICAL TRIAL: NCT05609981
Title: Optimising Medication With Focus on Deprescribing in Frail Older People With Multidose Drug
Brief Title: Optimising Medication With Focus on Deprescribing in Frail Older People With Multidose Drug Dispensing Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SIR Institute for Pharmacy Practice and Policy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UPF2211; 80-86600-98-19512 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Deprescriptions; Polypharmacy; Primary Health Care; Community Pharmacy Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Other): The intervention at t=0 consists of a 5-step patient-centred CMR focused on deprescribing supported by a toolbox provided to the pharmacists
  Interventions: Other: Clinical medication review focused on deprescribing
- Control (No Intervention): Usual care.

INTERVENTIONS:
Other: Clinical medication review focused on deprescribing — A pharmacist-led intervention consisting of a clinical medication review with the focus on deprescribing in older patients using multidose drug dispensing (MDD) systems.
  Pharmacist are trained in deprescribing and a developed toolbox to support the intervention is provided
  Arms: Intervention

SUMMARY:
Overuse is common in frail older people with polypharmacy, especially in frail older users of multidose drug dispensing (MDD) systems. In this study, we will investigate the effect of a clinical medication review (CMR) with integration of deprescribing (toolbox) on the number of ceased and dose lowered medications (persistent after 6 months) compared to usual care in older users of MDD systems with hyperpolypharmacy.

We will perform a controlled cluster-randomized trial in 38 community pharmacies. Per pharmacy, 10 older patients (>= 75) with hyperpolyfpharmacy (>10 medicines in use) with a MDD will be included. Pharmacists will receive training to perform the intervention, a 5-step CMR with a deprescribing toolbox (including deprescribing protocols): 1) patient interview; 2) pharmacotherapeutic analysis; 3) pharmacist and GP discuss actions; 4) actions are discussed with patient; 5) (two)weekly follow-up.

DETAILED DESCRIPTION:
AIM: is to investigate the effect of a clinical medication review in combination with a toolbox about deprescribing.

STUDY DESIGN: a controlled cluster-randomized trial will be performed, in which participating pharmacists in the Netherlands will be randomized to conduct clinical medication reviews with 10 eligible patients (intervention) or to provide usual care (control).

STUDY POPULATION: hyperpolypharmacy (≥ 10 chronic drugs) older patients (≥75 years) using a multidose drug dispensing (MDD) system

INTERVENTION: the intervention at t=0 consists of a 5-step patient-centred CMR focuses on deprescribing supported by the toolbox developed in WP1. The CMR starts with a patient interview (step 1) by a community pharmacist focussing on patient's preferences with input from the questionnaires on healthproblems, frailty and patient wishes. After the pharmacotherapeutic analysis (step 2), the pharmacist and the GP discuss the identified patient preferences and possible actions, including deprescribing (step 3). When patients are treated for one of more disease by a hospital specialist, pharmacist or GP consults this physician when appropriate. The health care providers decide together with the patient which actions will be conducted and their priority. This will result in a pharmaceutical care plan taking into account the tapering schemes from the deprescribing protocols (step 4). All actions and deprescribing steps will be evaluated with the patient during at least two follow-up moments (or more according to the patient's needs) to monitor the results of the actions. The follow-up moments can be performed by nurse practitioners or GPs with consultation of the community pharmacist when needed, e.g. to adapt tapering schemes based on the patient's health problems or withdrawal symptoms (step 5).

CONTROL: usual care.

OUTCOME MEASURES: the primary outcome measure is the number of ceased or dose lowered drugs per patient persistent after 6 months. Secondary, PREMs and PROMs including quality of life will be measured, as well as intermediate outcomes and process related outcomes

DATA-ANALYSIS: Intention-to-treat analysis and a per-protocol-analysis for the primary outcome and PROM, and an explorative subgroup analysis (age, gender, health problems, number of medicines in use). Descriptive analysis of other outcomes (intervention group only).

SAMPLE SIZE: To detect an effect size of 1 ceased / dose lowered drug (standard deviation 2.5), 80% power and α=0.05, we need a total of 266 patients for the analysis of the primary outcome and to account for clustering effects within pharmacies (ICC = 0,05 and clustersize = 7). Taking loss to follow-up into account (35%), 38 teams need to recruit 10 patients each.

ELIGIBILITY:
Inclusion Criteria:

* using a multidose drug dispensing system
* hyperpolypharmacy patient (using 10 drugs or more)
* age: 75 years or older

Exclusion Criteria:

* received a CMR in the previous 12 months
* incapacitated
* patients for whom the general practitioner is not the primary practionar
* expected lifespan of less than six motnhs
* patients who live in a nursing home

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 318 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
number of ceased or dose lowered drugs per patient | 6 months after the start of the medication review (t = 6 months)
  number of ceased or dose lowered drugs per patient based on dispensing data

CONTACTS AND LOCATIONS:
Locations (1):
- SIR Institute for Pharmacy Practice and Policy, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided